CLINICAL TRIAL: NCT06673121
Title: Respiratory Disease Cohort Studies of Chinese Medicine for Pulmonary Nodule （RESEARCH-PN）
Brief Title: Respiratory Disease Cohort Studies of Chinese Medicine for Pulmonary Nodule
Status: Recruiting | Type: Observational
Sponsor: Third Affiliated Hospital of Henan University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: RESEARCH-Pulmonary nodule
Record Dates: First submitted 2024-09-26; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-09

CONDITIONS: Pulmonary Nodule; Cohort Study; Traditional Chinese Medicine
Keywords: Pulmonary nodule; Cohort study; Traditional Chinese Medicine
MeSH Terms: interventions — Medicine, Chinese Traditional

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Traditional Chinese Medicine Group: Patients with pulmonary nodules treated with traditional Chinese medicine
  Interventions: Drug: Traditional Chinese Medicine
- Non-Traditional Chinese Medicine Treatment Group: Patients with pulmonary nodules have not received traditional Chinese medicine treatment

INTERVENTIONS:
Drug: Traditional Chinese Medicine — Received treatment with traditional Chinese medicine
  Groups: Traditional Chinese Medicine Group

SUMMARY:
This study is a prospective multicenter cohort study that primarily evaluates the impact of traditional Chinese medicine treatment on pulmonary nodules

DETAILED DESCRIPTION:
This study is a multicenter, prospective cohort study that will recruit at least 2244 individuals with chest HRCT findings of pulmonary nodules and recommended follow-up by MDT from four research centers. According to whether patients with pulmonary nodules are treated with traditional Chinese medicine, they are divided into a traditional Chinese medicine cohort and a non-traditional Chinese medicine cohort , and are followed up for at least 2 years. The main outcome measures were pulmonary nodule growth (enlargement or new onset) and nodule regression (reduction or disappearance). To evaluate the efficacy of traditional Chinese medicine treatment for patients with pulmonary nodules, secondary outcome measures include nodule volume, average nodule density, doubling time of volume, internal and external signs of nodules, anxiety self-assessment scale, depression self-assessment scale and SF-36 scale.

ELIGIBILITY:
Inclusion Criteria:

① Patients with pulmonary nodules and recommended for follow-up by MDT; ② Voluntarily sign the informed consent form.

Exclusion Criteria:

①Patients with metastatic pulmonary nodules; ②Patients with benign diseases such as pulmonary lymph nodes, hamartomas, sclerosing alveolar cell tumors, or nodules with obvious benign features such as calcification; ③Patients withserious heart, lung, liver and kidney diseases.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with pulmonary nodules have no age or gender restrictions
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Pulmonary nodule growth | Low risk pulmonary nodules measure at month 12, 24,36,48 and60. Medium risk pulmonary nodules measure at month 6,12,18,24,30,36,42,48,54and 60. High risk pulmonary nodules measure at 3,6,9,12,15,18,21,24,27,30, 33,36,39,42,45,48,51,54,57 and 60.
  Enlargement of pulmonary nodules or appearance of new pulmonary nodules
Pulmonary nodule regression | Low risk pulmonary nodules measure at month 12, 24,36,48 and60. Medium risk pulmonary nodules measure at month 6,12,18,24,30,36,42,48,54and 60. High risk pulmonary nodules measure at 3,6,9,12,15,18,21,24,27,30, 33,36,39,42,45,48,51,54,57 and 60.
  Shrinkage or disappearance of pulmonary nodules

SECONDARY OUTCOMES:
Nodule stability | Low risk pulmonary nodules measure at month 12, 24,36,48 and60. Medium risk pulmonary nodules measure at month 6,12,18,24,30,36,42,48,54and 60. High risk pulmonary nodules measure at 3,6,9,12,15,18,21,24,27,30, 33,36,39,42,45,48,51,54,57 and 60.
  The volume change of pulmonary nodules is within ± 15%
Pulmonary nodule volume | Low risk pulmonary nodules measure at month 12, 24,36,48 and60. Medium risk pulmonary nodules measure at month 6,12,18,24,30,36,42,48,54and 60. High risk pulmonary nodules measure at 3,6,9,12,15,18,21,24,27,30, 33,36,39,42,45,48,51,54,57 and 60.
  Calculate through chest HRCT and AI analysis
Mean density of pulmonary nodules | Low risk pulmonary nodules measure at month 12, 24,36,48 and60. Medium risk pulmonary nodules measure at month 6,12,18,24,30,36,42,48,54and 60. High risk pulmonary nodules measure at 3,6,9,12,15,18,21,24,27,30, 33,36,39,42,45,48,51,54,57 and 60.
  Calculate through chest HRCT and AI analysis
Doubling time of pulmonary nodule volume | Low risk pulmonary nodules measure at month 12, 24,36,48 and60. Medium risk pulmonary nodules measure at month 6,12,18,24,30,36,42,48,54and 60. High risk pulmonary nodules measure at 3,6,9,12,15,18,21,24,27,30, 33,36,39,42,45,48,51,54,57 and 60.
  Through AI analysis and calculation
Internal signs of pulmonary nodules | Low risk pulmonary nodules measure at month 12, 24,36,48 and60. Medium risk pulmonary nodules measure at month 6,12,18,24,30,36,42,48,54and 60. High risk pulmonary nodules measure at 3,6,9,12,15,18,21,24,27,30, 33,36,39,42,45,48,51,54,57 and 60.
  The HRCT manifestations of pulmonary nodules include vacuolar sign, bronchial sign, cystic sign, microvascular sign, etc
External signs of pulmonary nodules | Low risk pulmonary nodules measure at month 12, 24,36,48 and60. Medium risk pulmonary nodules measure at month 6,12,18,24,30,36,42,48,54and 60. High risk pulmonary nodules measure at 3,6,9,12,15,18,21,24,27,30, 33,36,39,42,45,48,51,54,57 and 60.
  The external features of pulmonary nodules include morphology, boundaries, margins, spicules, pleural traction, etc
self-rating anxiety scale | Scale will be measured at 3,6,9,12,15,18,21,24,27,30, 33,36,39,42,45,48,51,54,57 and 60. A score of 50-59 is defined as mild anxiety, and 60-69 is defined as moderate anxiety , and a score of 70 or above is defined as severe anxiety.
  Evaluate the anxiety status of patients with pulmonary nodules
self-rating depression scale | Scale will be measured at 3,6,9,12,15,18,21,24,27,30, 33,36,39,42,45,48,51,54,57 and 60. A score of ≥ 53 indicates the presence of depression.
  Evaluate the depression status of patients with pulmonary nodules
SF-36 scale | Scale will be measured at 3,6,9,12,15,18,21,24,27,30, 33,36,39,42,45,48,51,54,57 and 60.The scores in all aspects are from 0 to 100 points, and the higher the score, the better the quality of life.
  Evaluate the quality of life of patients with pulmonary nodules

CONTACTS AND LOCATIONS:
Overall Officials: Jiansheng LI, Professor, Study Chair — The First Affiliated Hospital of Henan University of Traditional Chinese Medicine
Locations (1):
- The Third Affiliated Hospital of Henan University of Traditional Chinese Medicine, Zhengzhou, Henan, China